CLINICAL TRIAL: NCT04089111
Title: Does Automatically Generated Tidal Volumes With Closed-loop Ventilation Leads to Safe Transpulmonary Pressures in Intubated Chronic Obstructive Pulmonary Disease Patients?
Brief Title: Closed Loop Ventilation With High Tidal Volumes and Safe Transpulmonary Pressure in COPD (COPD-SAFE)
Acronym: COPD-SAFE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Cenk Kirakli, M.D., Associate Professor Cenk Kirakli. M.D., Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: IGHCEAH-ICU-4
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Mechanical ventilation; Adaptive Support Ventilation; Transpulmonary pressure; Intrinsic PEEP; Safety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Positive-Pressure Respiration, Intrinsic

STUDY DESIGN:
Intervention Model Description: Patients will be ventilated for two different minute volume targets in two sets. 'Adapted support ventilation' and 'volume control (VC)' modes will be used consecutively in each set. Every patient will be ventilated 1.1. ASV with minute volume target of % 100; 1.2. VC with same MV target; 2.1 ASV with MV target associated with PaCo2 less than 45 mmHg; 2.2 VC with same MV target. Sequence of ventilation modes wıll be randomized within each group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be aware of the procedure or ventilation modes that will be performed. Outcomes will be analyzed by an independent statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1.1. ASV, MV target 100% (Experimental): Patients will be ventilated with ASV mode. Tidal volume, ventilation frequency, inspiratory duration will be automatically adjusted by the mechanical ventilator.
  Interventions: Other: Minute volume target of 100%
- 1.2. Volume control, MV target %100 (Active Comparator): Patients will be ventilated with volume control mode. A tidal volume of 6-8 ml/kg will be used. I:E ratio will be set as 1:3 Ventilation frequency will be adjusted to reach the same volume target calculated in arm1.
  Interventions: Other: Minute volume target of 100%
- 2.1. ASV, MV target to reach PaCO2< 45 mmHg (Experimental): Patients will be ventilated with ASV mode. Tidal volume, ventilation frequency, inspiratory duration will be automatically adjusted by the mechanical ventilator.
  Interventions: Other: Minute volume target to reach PaCO2 less than 45% (high tidal volume)
- 2.2. Volume control, MV target to reach PaCO2< 45 mmHg (Active Comparator): Patients will be ventilated with volume control mode. A tidal volume of 6-8 ml/kg will be used. I:E ratio will be set as 1:3. Ventilation frequency will be adjusted to reach the target PaCO2 level
  Interventions: Other: Minute volume target to reach PaCO2 less than 45% (high tidal volume)

INTERVENTIONS:
Other: Minute volume target of 100% — Patients will be ventilated to reach minute volume target of %100 (100 ml per ideal body weight).
  Arms: 1.1. ASV, MV target 100%; 1.2. Volume control, MV target %100
Other: Minute volume target to reach PaCO2 less than 45% (high tidal volume) — Patients will be ventilated to reach minute volume target associated with PaCO2 less than 45%.
  Arms: 2.1. ASV, MV target to reach PaCO2< 45 mmHg; 2.2. Volume control, MV target to reach PaCO2< 45 mmHg

SUMMARY:
This study evaluates the safety and efficacy of high tidal volumes generated by "Adapted Support Ventilation (ASV) mode' in mechanically ventilated severe COPD patients. Every patient will be ventilated consecutively with ASV and Volume Control (VC) modes at 2 different levels of minute volume in 2 sets. ASV mode is expected to be safe measured by adequate inspiratory transpulmonary pressures and expected to be as effective as VC mode with lower intrinsic positive end expiratory pressure (iPEEP) levels.

DETAILED DESCRIPTION:
Acute exacerbations of Chronic Obstructive Pulmonary Disease (COPD) may require mechanical ventilation. Various mechanical ventilation strategies and modes can be used to manage respiratory insufficiency in such patients. High tidal volumes required for mechanical ventilation of patients with obstructive pathologies is a well-known fact. Adapted Support Ventilation (ASV) is an intelligent closed-loop mechanical ventilation mode which automatically adjusts ventilation to lung mechanics. Led by measured lung mechanics, ASV mode often generates higher than usual tidal volumes during mechanical ventilation of COPD patients, particularly if the minute volume (MV) target is high. Thus, the effects of high tidal volumes on inspiratory transpulmonary pressure (Ptp), and whether Ptp stays within safe limits during ASV mode is of great interest.

Patients with acute exacerbation of COPD who required mechanical ventilation will be enrolled in the first 24 hours of admission to the intensive care unit. All patients will be deeply sedated. An esophageal balloon catheter will be inserted in order to measure transpulmonary pressure. 100 % minute volume target will be calculated in advance as 100 ml per ideal body weight.

Patients will be ventilated with two different MV targets in two sets. 'Adapted support ventilation' and 'volume control (VC)' modes will be used consecutively within each set. While the target minute volume will be 100 % in the first set, the volume target in the second set will be tuned to decrease patients PaCO2 below 45 mmHg. The sequence of ventilation mode will be randomized within each set. Ventilation periods will be 30 minutes with 15 minutes washout period in between. İf Ptp increase above 20 cmH20 at any ventilation mode, the tidal volume will be decreased.

ASV mode is expected to be safe, assessed by adequate inspiratory transpulmonary pressures, and expected to be as effective as VC mode with lower intrinsic positive end expiratory pressure (iPEEP) levels.

ELIGIBILITY:
Inclusion Criteria:

* Acute exacerbation of Chronic Obstructive Lung Disease
* Being intubated for less than 24 hours
* Not being planned to be extubated in 24 hours
* Expiratory time constant (RCexp) more than > 2.0 s

Exclusion Criteria:

* Restrictive lung pathologies
* Impaired hemodynamic status
* Esophageal pathologies
* Bronchopleural fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Transpulmonary inspiratory pressure (Ptinsp) | 30'th minute of each intervention arm
  Ptpinsp will be measured with an inspiratory pause maneuver.

SECONDARY OUTCOMES:
Intrinsic Positive End Expiratory Pressure (PEEPi) | 30'th minute of each intervention arm
  PEEPi will be measured with an expiratory hold maneuver.

OTHER OUTCOMES:
Mean arterial pressure | 30'th minute of each intervention arm
  Mean arterial pressure measured by invasive or non-invasive methods
PaO2, FiO2 ratio | 30'th minute of each intervention arm
  Ratio of arterial partial oxygen pressure to inspired fraction of oxygen
Heart rate | 30'th minute of each intervention arm
  Heart rate measured by ECG

CONTACTS AND LOCATIONS:
Overall Officials: Sami C Kirakli, MD, Principal Investigator — Dr. Suat Seren Chest Diseases and Surgery Educatin and Resarch Hospital
Locations (1):
- Izmir Dr. Suat Seren Chest Diseases and Surgery Education and Research Hospital, Intensive Care Unit, Izmir, Yenisehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507
- [Background] Grieco DL, Chen L, Brochard L. Transpulmonary pressure: importance and limits. Ann Transl Med. 2017 Jul;5(14):285. doi: 10.21037/atm.2017.07.22. PMID 28828360
- [Background] Mauri T, Yoshida T, Bellani G, Goligher EC, Carteaux G, Rittayamai N, Mojoli F, Chiumello D, Piquilloud L, Grasso S, Jubran A, Laghi F, Magder S, Pesenti A, Loring S, Gattinoni L, Talmor D, Blanch L, Amato M, Chen L, Brochard L, Mancebo J; PLeUral pressure working Group (PLUG-Acute Respiratory Failure section of the European Society of Intensive Care Medicine). Esophageal and transpulmonary pressure in the clinical setting: meaning, usefulness and perspectives. Intensive Care Med. 2016 Sep;42(9):1360-73. doi: 10.1007/s00134-016-4400-x. Epub 2016 Jun 22. PMID 27334266
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647